CLINICAL TRIAL: NCT02280824
Title: Transcaval Access for Transcatheter Aortic Valve Replacement in Patients With No Good Options for Aortic Access
Brief Title: Transcaval Access for Transcatheter Aortic Valve Replacement in People With No Good Options for Aortic Access
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999915009; 15-H-N009
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-12-28

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcaval; TAVR; AMPLATZER(R) Occluder
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- A (Experimental): Transcaval acesss for transcatheter aortic valve replacement in patients with no good options for aortic access
  Interventions: Procedure: CA-TAVR; Device: Amplatzer Duct Occluder

INTERVENTIONS:
Procedure: CA-TAVR — Transcaval acesss for transcatheter aortic valve replacement in patients with no good options for aortic access
Device: Amplatzer Duct Occluder

SUMMARY:
Background:

- Some people who need a transcatheter aortic valve replacement (TAVR) have leg arteries that are too small and are too sick for standard techniques. But they may benefit from a new technique called transcaval TAVR. For this technique, doctors make a hole between the largest vein (vena cava) and largest artery (aorta) in the body, inside the abdomen. Then they replace the valve through a tube they put in the groin vein. Then they close the hole between the vein and the artery using a device designed to close holes in the heart. This study tests the device for this new, off-label use.

Objective:

- To further study the safety and effectiveness of transcaval TAVR.

Eligibility:

- Adults age 21 and older who would benefit from TAVR but for whom standard techniques are not suitable.

Design:

* Participants will be selected by a team of heart specialists and others.
* Participants will have a computed tomography (CT) scan with or without contrast dye.
* Participants will have blood tests.
* Participants will have transcaval TAVR.
* Participants will receive the same standard care as for all patients with TAVR.
* Participants will also have another CT scan, or an MRI or ultrasound, before they leave the hospital, and again after about 30 days and after about 12 months.
* Participants will be contacted 1 and 6 months afterwards and will have another visit 1 year later. They will have a CT, MRI, or ultrasound. They will have blood tests and a physical exam.

DETAILED DESCRIPTION:
Transcaval access to the abdominal aorta from the neighboring inferior vena cava (IVC) has enabled transcatheter aortic valve replacement (TAVR) in a small number of patients who have no good options for standard percutaneous femoral access or for standard surgical access to the cardiac apex or to the ascending aorta. In this prospective registry we will collect data from multiple medical centers as they offer transcaval TAVR to patients with extreme or prohibitive risk of conventional TAVR.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults age greater than or equal to 21 years
* Severe symptomatic de novo aortic valve stenosis or bioprosthetic aortic valve failure for which transcatheter aortic valve replacement (TAVR) is felt beneficial according to the consensus of the institutional multidisciplinary heart team
* Extreme risk or inoperability for TAVR via conventional femoral artery, trans-apical, or trans-aortic access in the determination of the multidisciplinary heart team. This determination includes an in-person consultation by at least one cardiac surgeon member of the heart team.
* Anatomic eligibility for caval-aortic TAVR, graded as favorable or feasible based on NHLBI core lab assessment of the baseline CT examination.

EXCLUSION CRITERIA:

* Unable or unwilling to consent to participate
* Anatomic eligibility for caval-aortic TAVR graded as unfavorable based on NHLBI core lab assessment of the baseline CT examination
* Unlikely to benefit from caval-aortic TAVR
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-10-30; Primary Completion 2017-07-27 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is device success, which is defined as successful transcaval access and deployment of a closure device without death or emergency open surgery related to caval-aortic access | 1 year
  The primary endpoint is device success, which is defined as successful transcaval access and deployment of a closure device without death or emergency open surgery related to caval-aortic access

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (15):
- United States (15):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston Hospital, Evanston, Illinois
  - Advocate Heart Institute, Oakbrook Terrace, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - York Hospital, York, Pennsylvania
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - University of Virginia Medical Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Medical Center, Roanoke, Virginia

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Greenbaum AB, O'Neill WW, Paone G, Guerrero ME, Wyman JF, Cooper RL, Lederman RJ. Caval-aortic access to allow transcatheter aortic valve replacement in otherwise ineligible patients: initial human experience. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2795-804. doi: 10.1016/j.jacc.2014.04.015. Epub 2014 May 7. PMID 24814495
- [Background] Halabi M, Ratnayaka K, Faranesh AZ, Chen MY, Schenke WH, Lederman RJ. Aortic access from the vena cava for large caliber transcatheter cardiovascular interventions: pre-clinical validation. J Am Coll Cardiol. 2013 Apr 23;61(16):1745-6. doi: 10.1016/j.jacc.2013.01.057. Epub 2013 Apr 2. No abstract available. PMID 23500317
- [Derived] Lederman RJ, Babaliaros VC, Rogers T, Stine AM, Chen MY, Muhammad KI, Leonardi RA, Paone G, Khan JM, Leshnower BG, Thourani VH, Tian X, Greenbaum AB. The Fate of Transcaval Access Tracts: 12-Month Results of the Prospective NHLBI Transcaval Transcatheter Aortic Valve Replacement Study. JACC Cardiovasc Interv. 2019 Mar 11;12(5):448-456. doi: 10.1016/j.jcin.2018.11.035. PMID 30846083
- [Derived] Greenbaum AB, Babaliaros VC, Chen MY, Stine AM, Rogers T, O'Neill WW, Paone G, Thourani VH, Muhammad KI, Leonardi RA, Ramee S, Troendle JF, Lederman RJ. Transcaval Access and Closure for Transcatheter Aortic Valve Replacement: A Prospective Investigation. J Am Coll Cardiol. 2017 Feb 7;69(5):511-521. doi: 10.1016/j.jacc.2016.10.024. Epub 2016 Oct 29. PMID 27989885